CLINICAL TRIAL: NCT02966717
Title: The Clinical Study of Rituximab Combined With Mesenchymal Stem Cells in the Treatment of Primary Nephrotic Syndrome (3-4 Stage of Chronic Kidney Disease)
Brief Title: Rituximab Combined With MSCs in the Treatment of PNS (3-4 Stage of CKD)
Acronym: CKD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tangxun8022
Record Dates: First submitted 2016-10-30; First posted 2016-11-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Renal Insufficiency, Chronic; Nephrotic Syndrome
Keywords: Rituximab; Mesenchymal stem cells; primary nephrotic syndrome; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parallel control of conventional therapy (Active Comparator): Intervention of conventional therapy group: controlling blood pressure using amlodipine, valsartan, metoprolol and terazosin and so on , protecting the renal function using bailing capsule, alpha keto acid, low molecular weight heparin and so on.
  Interventions: Drug: conventional therapy
- experimental group (Experimental): Intervention of Rituximab combined with mesenchymal stem cells group: as follows, Rituximab, 100mg/time every one week, the infusion should be a total of 4 times; and then after at least 4 days interval after the first and the third infusion of the Rituximab , the dosage of mesenchymal stem cells tends to be 10^6/kg/time every 2 weeks, while the infusion should be a total of 2 times.
  Interventions: Drug: Rituximab; Drug: Mesenchymal stem cells

INTERVENTIONS:
Drug: Rituximab — Rituximab is a human-mouse-chimeric monoclonal antibody which was approved in 1997 for the treatment of cancer.
  Other Names: Mabthera; RTX; Rituxan
  Arms: experimental group
Drug: conventional therapy — Intervention of conventional therapy group: controlling blood pressure using amlodipine, valsartan, metoprolol and terazosin and so on , protecting the renal function using bailing capsule, alpha keto acid, low molecular weight heparin and so on.
  Arms: parallel control of conventional therapy
Drug: Mesenchymal stem cells — Mesenchymal stem cells (MSCs), which belongs to mesoderm, is a kind of somatic stem cell with the ability of self-replication and the potential of multi-directional differentiation.
  Other Names: MSCs
  Arms: experimental group

SUMMARY:
Primary nephrotic syndrome(PNS) is a group of clinical symptoms caused by a variety of factors, including immune,environmental, genetic, et al. Oral corticosteroids have been to be the preferred drug for the treatment of PNS, but the long-term use of glucocorticoid therapy in clinic often induces some problems such as hormone dependent and hormone resistance, as well as severe side effects which act as a threat to the patients' health. Besides, patients with proteinuria long-term not control often behave faster progression into chronic renal failure, leading to poor prognosis. In renal diseases, Rituximab ( RTX) is often used in the treatment of refractory nephropathy, such as hormone dependent nephrotic syndrome, hormone resistance nephrotic syndrome, frequency recurrence nephrotic syndrome, which shows exciting effects in delaying the development of the disease.At present, mesenchymal stem cells ( MSCs) has been used as a research hotspot to repair the tissue damage of chronic kidney disease, and it also behaves certain effects. The purpose of this study is to seek a more targeted treatment, more precise curative effect and more feasibility treatment for PNS(CKD3-4),so as to delay or reverse the disease and improve the quality of life of patients with CKD.

DETAILED DESCRIPTION:
Primary nephrotic syndrome(PNS) is a group of clinical symptoms caused by a variety of factors, including immune,environmental, genetic, et al. Oral corticosteroids have been to be the preferred drug for the treatment of PNS, but the long-term use of glucocorticoid therapy in clinic often induces some problems such as hormone dependent and hormone resistance, as well as severe side effects which act as a threat to the patients' health. On the treatment of nephrotic syndrome in the latest evidence-based practice guidelines, Japan and Kidney Disease: Improving Global Outcomes(KDIGO) still have no high-level-evidence recommendation for the steroid resistant PNS and those patients with renal function significantly impaired. In addition, a large number of patients with proteinuria long-term not control often behave faster progression into chronic renal failure, leading to poor prognosis. What's more, patients holding the progression into 3-4 stage of chronic kidney disease with nephrotic syndrome ofen can not tolerate the conventional immunosuppressive therapy, thus cause faster progression into end-stage renal disease. There is no better treatment method for this phenomenon nowadays. Therefore, it is particularly important to explore new treatment options for the clinical disease described above.

In renal diseases, Rituximab ( RTX) is often used in the treatment of refractory nephropathy, such as hormone dependent nephrotic syndrome, hormone resistance nephrotic syndrome, frequency recurrence nephrotic syndrome, which shows exciting effects in delaying the development of the disease. An observational、 multicenter、 retrospective study about the therapeutic effect of RTX on adult minimal change nephrotic syndrome (MCNS) was conducted. This study confirmed that RTX is safe and effective in the treatment of adult patients with MCNS, which can be used as an alternative treatment options for MCNS patients with long-term recurrence. Whereas, whether the rituximab in the treatment of PNS (MCNS or other types of NS) combined with CKD plays the same role on delaying the progression of renal disease, there is no relevant clinical trials reported.

At present, mesenchymal stem cells ( MSCs) has been used as a research hotspot to repair the tissue damage of chronic kidney disease, and it also behaves certain effects. Clinical Studies about the treatment of PNS by the umbilical cord mesenchymal stem cells or the treatment of CKD by the bone marrow mesenchymal stem cells suggest that the mesenchymal stem cells can improve the patients's condition with PNS or CKD. However, cell therapy in the clinical trials in patients with CKD is rarely to be seen, and there is no definitive conclusion. Accordingly, more clinical studies are needed to assess the effectiveness, feasibility and safety of cell therapy, as well as formulating standard treatment plans.

We have accumulated 3 cases of patients with chronic kidney disease(in the 3-4 stage), accompanied with a large number of proteinuria and renal function declining rapidly, providing RTX infusion combined with mesenchymal stem cell.

Of which, 3 patients had significantly reduced proteinuria, 2 cases showed different levels improvement of renal function, 1 cases kept stable renal function. There was no obvious adverse reaction and safety risk, but more clinical trials was still required. In addition, our team has carried out a project about autologous non-clearing bone marrow stem cell transplantation in the treatment of severe lupus associated with renal function impaired. This study revealed good treatment effect, which can provide some certain clinical work foundation and experience for our following research.

In summary, we intend to conduct a prospective、 single-center、 randomized 、controlled clinical study, uniting the Third Affiliated Hospital of Southern Medical University together to explore the effectiveness and safety of rituximab combined with mesenchymal stem cells for the treatment of PNS(CKD3-4). The purpose of this study is to seek a more targeted treatment, more precise curative effect and more feasibility treatment for PNS(CKD3-4),so as to delay or reverse the disease and improve the quality of life of patients with CKD.

ELIGIBILITY:
Gender-Definition: Physical gender of individuals who may participate in the protocol. Select one-Both: both female and male participants are being studied.

Age Limits-Minimum Age( Definition: Minimum age of participants. ); Maximum Age (Definition: Maximum age of participants).

Accepts Healthy Volunteers?-Definition: Indicate if persons who have not had the condition(s) being studied or otherwise related conditions or symptoms, as specified in the eligibility requirements, may participate in the study.

Eligibility Criteria-Definition: Summary criteria for participant selection. The preferred format includes lists of inclusion and exclusion criteria as shown below.

Inclusion Criteria: A. Nephrotic syndrome(urine protein > 3.5g/d and serum albumin < 30g/L）； B. 3-4 stage of CKD [glomerular filtration rate 15-59 ml/ (min ·1.73m²)]； C. Age should be 18-65 years old； D. Accept treatment and signe informed consent voluntarily.

- Exclusion Criteria:A. Secondary nephrotic syndrome such as systemic lupus erythematosis nephritis, anaphylactic purpura nephritis and diabetic nephropathy and so on； B. Complications like severe infection, cardiovascular diseases, severe heart and lung as well as liver complications； C. Dialysis is extremely urgent； D. Obstructive urinary tract diseases； E. Creatinine rises more than 30% of the based value in nearly 3 months； F. Pregnancy or in lactation； G. Any other conditions that researchers consider not suitable to participate in this trial.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The change of serum creatinine elevation | 4 weeks, 8 weeks, 12 weeks
  The serum creatine elevation should be tested for at least 4 times, as follows, before treatment, 4 weeks after treatment, 8 weeks after treatment, 12 weeks after treatment.
The percentage of end-stage renal disease or death. | 3 years
  The percentage of end-stage renal disease or death should be less than 60%.

CONTACTS AND LOCATIONS:
Overall Officials: Tang Xun, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided